CLINICAL TRIAL: NCT00744445
Title: Erythropoietin Therapy in Patients With Chronic Renal Failure: A Study of Time Dependent Activity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Dr. G.A. Bjarnason, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 022-1994
Record Dates: First submitted 2008-08-29; First posted 2008-09-01 (Estimated); Last update posted 2008-09-01 (Estimated); Status verified 2008-08

CONDITIONS: Hemodialysis; Chronic Renal Failure; Anemia
Keywords: hemodialysis; erythropoietin
MeSH Terms: conditions — Kidney Failure, Chronic; Anemia | interventions — Erythropoietin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 0800 (Active Comparator): r-HuEPO administered at 0800 hrs
  Interventions: Drug: r-HuEPO
- 1500 (Active Comparator): r-HuEPO administered at 1500 hrs
  Interventions: Drug: r-HuEPO
- 2200 (Active Comparator): r-HuEPO administered at 2200 hrs
  Interventions: Drug: r-HuEPO

INTERVENTIONS:
Drug: r-HuEPO — r-HuEPO 50 U/kg s.c. three times per week. The dose is rounded to the nearest 2000 unites.

SUMMARY:
The purpose of this research study was to determine if the activity of erythropoietin (r-HuEPO) is time dependent when given to chronic renal failure patients at three different times of day.

DETAILED DESCRIPTION:
This phase-II crossover study was designed to test if the activity of erythropoietin is time dependent. Patients with chronic renal failure on hemodialysis requiring r-HuEPO to maintain adequate levels of hematocrit are eligible for the study. Patients were administered r-HuEPO subcutaneously three times per week, 50 U/kg, rounded to the nearest 2000 units. r-HuEPO will be administered until the hematocrit rises from the baseline level of 20-24% to the target level of 30-34%. This will be repeated three times, each at different times of day, either 0800, 1500 or 2200 hrs and the order of these will be randomly determined. Each patient will complete all three of the phases.

ELIGIBILITY:
Inclusion Criteria:

* Chronic renal failure patients requiring hemodialysis and requiring r-HuEPO to maintain adequate hematocrit levels
* Serum ferritin level > 200 micrograms/L and transferrin saturation > 15%
* Serum erythropoietin level less than 500 mu/ml (when off r-HuEPO)
* Prior therapy with r-HuEPO
* An adequate program of dialysis established
* Informed consent signed

Exclusion Criteria:

* Adocumented cause of anemia other than chronic renal disease
* Symptoms of unstable coronary artery disease
* Poorly controled hypertension
* Known seizure disorder
* Other active inflammatory or infective disorders
* Other disorders that may diminish the response of the bone marrow to r-HuEPO

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 1993-10; Primary Completion 1998-08 (Actual); Study Completion 1998-08 (Actual)

PRIMARY OUTCOMES:
Time for hematocrit to rise

CONTACTS AND LOCATIONS:
Overall Officials: Georg Bjarnason, MD, FRCPC, Principal Investigator — Sunnybrook Health Sciences Centre